CLINICAL TRIAL: NCT02489396
Title: Promoting Healthier Food Purchases By Leveraging the Online-Grocery Environment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Lizzy Pope, Assistant Professor and DPD Director, University of Vermont
Other Study IDs: 029898
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Color

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Grocery Customers: All customers who shop on the Rosie site during the intervention period.
  Interventions: Behavioral: Nutrition facts automatically or not automatically displayed; Behavioral: Nutrition facts in color; Behavioral: Nutrition Facts Label in Larger Font; Behavioral: Healthier Items First

INTERVENTIONS:
Behavioral: Nutrition facts automatically or not automatically displayed — For two months nutrition information on the Rosie site will be displayed in a "tab" that consumers can click on to display the nutrition facts panels of products. Investigators will use NuVal scores to determine the fifteen "healthiest," and fifteen "least healthy" items in six grocery categories; chips, cookies, cereal & breakfast, yogurt, ice cream, and frozen pizza. We will then compare the number of clicks on nutrition information for healthier versus less healthy items to determine if there's a possibility of willful ignorance coming into play when choosing to purchase less healthy items.
Behavioral: Nutrition facts in color — For two months the font on products' nutrition facts labels will be displayed in red or green. For this proof-of-concept intervention, the color of a label's display will be determined randomly, in order to gather a clearer picture of whether label color could be leveraged to influence product choice. Items in each grocery category will be randomly assigned to receive green or red labels during the intervention period, so 50% of products in each category have red nutrition facts labels, and 50% have green nutrition facts labels. We will then compare proportions of green to red items purchased during the intervention period with the proportion of those same items purchased during the baseline period, when all labels were in black font.
Behavioral: Nutrition Facts Label in Larger Font — For two months the serving size and calorie lines on the nutrition facts labels will be displayed in a larger font for every item on the Rosie site. Average calories in customer purchases will be quantified using purchase data, and the average calories for online-grocery orders during baseline and intervention periods will be compared.
Behavioral: Healthier Items First — For two months, instead of the product popularity default-display option in the online store, thirty healthier items will be displayed on the first page in each grocery category. All grocery categories where there is scoring variation between healthy and less-healthy options (i.e. cereal, chips, bakery, sauces, etc.) will be included in the intervention. The thirty-targeted healthy items will be identified using NuVal scores. NuVal scores will not actually be displayed as part of the shopping site, and will be used exclusively as a guide to systematically determine targeted items in each food category. The proportion of targeted healthy items purchased in each category versus non-targeted items purchased during the intervention will be compared to the proportion of targeted vs. non-targeted items purchased during the baseline period.

SUMMARY:
Rationale: Online-grocery shopping is predicted to be one of the "hottest" food trends of 2014, as national retailers such as Amazon, as well as start-up companies, venture into the e- commerce grocery sector. Importantly, the online-grocery environment could be uniquely manipulated to promote healthier food purchasing and help with weight control. Since consumers tend to choose items listed first on menus and buffet lines, the order of food products displayed on the grocer's website may impact purchasing. Furthermore, it's possible that in an online-grocery environment, nutrition information could be made more salient to consumers. For example, previous research has demonstrated that label color influences perceptions of the healthfulness of foods. The FDA also recently proposed a redesign of foods' nutrition facts panels, which would highlight calorie content in a larger font. Although implementing this label change on all food labels could take years, e-commerce sites could change the format of the nutritional information they display much more quickly.

Objectives: The proposed study intends to nudge consumers to make healthier grocery purchases through three distinct interventions: 1.) Manipulating the order of food items within grocery categories; 2.) Displaying product nutrition information in red or green; and 3.) Presenting calorie information in a larger font size. We propose to examine these concepts in adult consumers using a grocery e-commerce platform servicing socioeconomically and racially diverse communities in the northeastern U.S.

ELIGIBILITY:
Inclusion Criteria:

* Shopping on a Rosie grocery site

Exclusion Criteria:

* No exclusion criteria, all orders will be eligible

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All orders placed on any of the Rosie sites or apps in the study period will be included. No active recruiting of participants will take place, data will only be collected from existing Rosie customers. Participants will not be informed that manipulations are happening on the website, other than notices the company occasionally displays when they are revising features of the website. In order to determine whether any of the proposed "mindless" interventions actually work, it is imperative that consumer attention not be drawn to changes in the site. It is expected that 400-1000 orders per month will be included as part of the study during each two-month intervention period.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Food Purchasing of targeted items | Continuously throughout the intervention expected average of 52 weeks
  Company purchasing records will be used to track purchasing of items during the baseline period, as well as during the intervention periods, for the healthier items displayed first and nutrition-facts label interventions.
Click Rate of targeted food items | Continuously throughout the intervention expected average of 52 weeks
  We will tabulate a "click-rate" for each targeted product during the intervention periods and at baseline to determine whether consumers clicked on the nutrition facts panels more often for healthier versus less-healthy products, and if consumers clicked more often when calories were displayed in larger fonts or were listed in red/green. We will also be able to determine whether customers clicked more often on the targeted healthy items when they were listed first on the website in each category. Clicks for each item will be tabulated weekly and averaged over the intervention or baseline periods.
Nutrient Analysis of Food Purchased by consumers | Continuously throughout the intervention expected average of 52 weeks
  To determine whether average number of calories purchased changed when calories and serving sizes were displayed in larger fonts, we will use purchasing data to compare the average number of calories purchased in orders before the font change to the average number of calories purchased during the font change. Calories per item will be determined using the USDA database, which houses nutrition facts for all foods on the Rosie website.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Because the data is coming from a private business, we do not plan to share the data publicly.